CLINICAL TRIAL: NCT02070289
Title: A Phase 1 Double Blind (3rd Party Open) Randomized, Placebo Controlled, Dose Escalation Study To Investigate The Safety, Tolerability And Pharmacokinetics Of Repeat Doses Of Pf-06372865 In Subjects Aged 18-55 (Group 1) And 56-75 Years (Group 2)
Brief Title: A Study to Evaluate Safety, Toleration and Time Course of Plasma Concentration of Multiple Oral Doses of PF-06372865 in Healthy Subjects of Two AgeGroups, Aged 18-55 Years (Group 1) and Aged 56-75 Years (Group 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7431002
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Multiple dose; safety; tolerability; PK
MeSH Terms: interventions — PF-06372865

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1: Cohort 1 (Experimental)
  Interventions: Drug: PF-06372865; Drug: Placebo
- Group 1: Cohort 2 (Experimental)
  Interventions: Drug: PF-06372865; Drug: Placebo
- Group 1: Cohort 3 (Experimental)
  Interventions: Drug: PF-06372865; Drug: Placebo
- Group 2: Cohort 4 (Experimental)
  Interventions: Drug: PF-06372865; Drug: Placebo
- Group 1 or 2: Cohort 5 (Experimental)
  Interventions: Drug: PF-06372865; Drug: Placebo
- Group 1 or 2: Cohort 6 (Experimental)
  Interventions: Drug: PF-06372865

INTERVENTIONS:
Drug: PF-06372865 — Tablets, 2.5 mg BID, 14 days
  Arms: Group 1: Cohort 1
Drug: Placebo — Tablets, BID, 14 days
  Arms: Group 1: Cohort 1
Drug: PF-06372865 — Tablets, to be decided dose, BID or titration, 14 days
  Arms: Group 1: Cohort 2
Drug: Placebo — Tablets, BID or titration, 14 days
  Arms: Group 1: Cohort 2
Drug: PF-06372865 — Tablets, to be decided dose, BID or titration, 14 days
  Arms: Group 1: Cohort 3
Drug: Placebo — Tablets, BID or titration, 14 days
  Arms: Group 1: Cohort 3
Drug: PF-06372865 — Tablets, to be decided dose, BID or titration, 14 days
  Arms: Group 2: Cohort 4
Drug: Placebo — Tablets, BID or titration, 14 days
  Arms: Group 2: Cohort 4
Drug: PF-06372865 — Tablets, to be decided dose, BID or titration, 14 days
  Arms: Group 1 or 2: Cohort 5
Drug: Placebo — Tablets, BID or titration, 14 days
  Arms: Group 1 or 2: Cohort 5
Drug: PF-06372865 — Tablets, to be decided dose, BID or titration, 14 days
  Arms: Group 1 or 2: Cohort 6

SUMMARY:
The purpose of this study is to investigate safety, toleration and time course of plasma concentration of multiple oral doses of PF-06372865 for 14 days in healthy subjects of two age groups, 18-55 years (Group 1) and 56-75 years (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* For Group 1 specific: Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive at Screening. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory.
* For Group 2 specific: Male and/or female subjects of non-childbearing potential between the ages of 56 and 75 years, inclusive at Screening. Subjects must be in reasonably good health as determined by the Investigator based on a detailed medical history, full physical examination (including blood pressure and pulse rate measurement), 12-lead ECG and clinical laboratory tests. Subjects with mild, chronic, stable disease (eg, osteoarthritis) may be enrolled if deemed medically prudent by the Investigator. At least 50% of the subjects enrolled in these cohorts must be 60 years of age and above at Screening.
* For Group 2 specific: Subjects taking daily prescription or non-prescription medications for management of acceptable chronic medical conditions must be on a stable dose of these, as defined by non change in dose for the 3 months prior to the first dose of study medication and no planned changes during the conduct of the study.

Exclusion Criteria:

* For Group 1 specific: Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* For Group 2 specific : Evidence or history of unstable disease or moderate to severe conditions which would, in the Investigator's opinion, interfere with the study evaluations or impact on the safety of participating subjects, such as orthostatic hypotension.
* Subjects with history of sleep apnea
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 14 days
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 14 days
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431002&StudyName=A%20Study%20to%20Evaluate%20Safety%2C%20Toleration%20and%20Time%20Course%20of%20Plasma%20Concentration%20of%20Multiple%20Oral%20Doses%20of%20PF-06372865%20in%20Healthy%20Subj